CLINICAL TRIAL: NCT01630733
Title: A Multinational, Randomized, Open-Label Phase III Study of Custirsen (TV-1011/OGX-011) In Combination With Docetaxel Versus Docetaxel As A Second-Line Treatment In Patients With Advanced or Metastatic (Stage IV) Non-Small Cell Lung Cancer
Brief Title: A Multinational, Randomized, Open-Label Study of Custirsen In Patients With Advanced or Metastatic (Stage IV) Non-Small Cell Lung Cancer
Status: Unknown | Phase: Phase 3 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Achieve Life Sciences (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: TV1011-LC-303; 2012-002447-14 (EudraCT Number)
Record Dates: First submitted 2012-06-26; First posted 2012-06-28 (Estimated); Last update posted 2016-07-01 (Estimated); Status verified 2016-06

CONDITIONS: Non-Small Cell Lung Cancer
Keywords: Metastatic; Stage IV; Advanced; lung cancer
MeSH Terms: conditions — Carcinoma, Non-Small-Cell Lung; Neoplasm Metastasis; Lung Neoplasms | interventions — OGX-011; Docetaxel

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Custirsen + Docetaxel (Experimental): Custirsen: Three loading doses of custirsen 640mg IV over 2 hours administered in 5 to 9 days prior to Day 1 of Cycle 1, then custirsen 640 mg IV weekly every 21-day cycle Docetaxel: 75 mg/m2 IV over 1 hour on Day 1 of every 21-day cycle
  Interventions: Drug: Custirsen; Drug: Docetaxel
- Docetaxel (Active Comparator): Docetaxel: 75 mg/m2 IV over 1 hour on Day 1 of every 21-day cycle Continue treatment until disease progression, unacceptable toxicity, withdrawal of consent or protocol specified parameters to stop treatment.
  Interventions: Drug: Docetaxel

INTERVENTIONS:
Drug: Custirsen — Custirsen: Three loading doses of custirsen 640 mg IV over 2 hours administered in 5 to 9 days prior to Day 1 of Cycle 1, then custirsen 640 mg IV weekly every 21-day cycle
  Other Names: OGX-011; TV-1011
  Arms: Custirsen + Docetaxel
Drug: Docetaxel — Docetaxel: 75 mg/m2 IV over 1 hour on Day 1 of every 21-day cycle

SUMMARY:
The primary objective of the study is to compare overall survival of patients randomized to receiving custirsen in combination with docetaxel (Arm A) with patients randomized to receive docetaxel alone (Arm B).

ELIGIBILITY:
Inclusion Criteria:

1. Patients must have a histologically or cytologically confirmed, unresectable, advanced or metastatic (Stage IV per AJCC 7th edition TNM staging) NSCLC
2. Males or females ≥ 18 years of age at screening.
3. Life expectancy of > 12 weeks from screening, according to the investigator's assessment.
4. Patients must have received one prior line of platinum-based systemic anticancer therapy for advanced or metastatic NSCLC. Prior maintenance therapy is allowed and will be considered as the same line of therapy when continued at the end of a treatment regimen.
5. Patients must have documented radiological disease progression either during or after the first-line therapy.
6. Patients must have at least one measurable lesion per RECIST 1.1 criteria.
7. ECOG performance status of 0 or 1 at screening.
8. Have adequate values, bone marrow, renal and liver functions at screening as defined below:

   * Absolute neutrophil count (ANC) ≥ 1.5 x 109/L
   * Platelet count ≥ 100 x 109/L
   * Hemoglobin ≥ 9 g/dL
   * Serum creatinine ≤ 1.5 x upper limit of normal (ULN)
   * Total Bilirubin ≤ 1.0 x ULN (unless elevated secondary to benign conditions such as Gilbert's disease)
   * AST and ALT ≤ 1.5 x ULN
9. Resolution of any toxic effects of prior therapy to Grade ≤1 according to NCI CTCAE, version 4.0 (exception of alopecia and ≤ Grade 2 peripheral neuropathy).
10. Females of child-bearing potential must have negative serum pregnancy test within 72 hours before randomization.
11. Women of child-bearing potential will practice a highly effective method of birth control during and for 3 months after the chemotherapy/ custirsen last dose. Men of reproductive potential who are not surgically sterile must agree to abstain from sexual activity or use medically accepted and highly effective method of contraception during and for 6 months after the chemotherapy/custirsen last dose.
12. Patients must be willing and able to give written informed consent prior to any protocol-specific procedures being performed and comply with the protocol requirements for the duration of the study.

Exclusion Criteria:

1. Patients treated with any systemic anti-cancer therapy for NSCLC within 21 days prior to randomization (6 weeks for Bevacizumab).
2. Radiotherapy ≤ 2 weeks prior to randomization. Patients must have recovered from all radiotherapy-related toxicities.
3. Major surgical procedure within 4 weeks prior to randomization. Patient must have recovered from all surgery-related complications.
4. Patients with known CNS metastases (Patients with any clinical signs of CNS metastases must have a CT or MRI of the brain to rule out CNS metastases in order to be eligible for participation in the study). Patients who have had brain metastases treated with radiotherapy or surgically removed with no residual disease confirmed by imaging; patients should be clinically stable and off corticosteroid treatment at least 3 weeks prior to randomization).
5. Patients with current diagnosis or a history of another active primary malignancy (except in situ carcinoma of the cervix, adequately treated non-melanomatous skin cancers, clinically localized prostate cancer, superficial bladder cancer or other malignancy treated at least 5 years previously with no evidence of recurrence).
6. Severe or unstable medical conditions such as heart failure, ischemic heart disease, uncontrolled hypertension, uncontrolled diabetes mellitus, psychiatric condition, as well as an ongoing cardiac arrhythmia requiring medication (≥ Grade 2, according to NCI CTCAE v4.0) or any other significant or unstable concurrent medical illness that in the opinion of the Investigator would preclude protocol therapy.
7. A history of events such as myocardial infarction, cerebrovascular accident or acute hepatitis within 3 months of randomization or treatment of a major active infection within one month of randomization, or any other significant event that in the opinion of the Investigator would preclude protocol therapy.
8. Planned concomitant participation in another clinical trial of an experimental agent, vaccine, or device. Concomitant participation in observational studies is acceptable.
9. Female patients who are breastfeeding.
10. Patients previously treated with docetaxel for NSCLC or with known severe hypersensitivity to taxane therapies.
11. Patients with known and documented EGFR mutation who have not received an EGFR inhibitor.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 700 (Estimated)
Dates: Start 2012-09; Primary Completion 2017-07 (Estimated); Study Completion 2017-07 (Estimated)

PRIMARY OUTCOMES:
Overall Survival | 60 months
  Primary endpoint and variable for the study is overall survival (OS), defined as the time from date of randomization to the date of death from any cause.

SECONDARY OUTCOMES:
Progression Free Survival per RECIST v1.1 | 60 months
  Progression Free Survival: time from date of randomization to first objective documented progression per Response Evaluation Criteria In Solid Tumors (RECIST) v1.1 or death due to any cause, whichever occurs first. Tumor lesions measured in at least one dimension with minimum size of 10 mm by CT scan, 10 mm caliper by clinical exam. Malignant lymph nodes must be >15 mm in short axis when assessed by CT scan. All measurable lesions up to a maximum of 2 lesions per organ and 5 in total representative of all involved organs should be identified as target lesions and measured and recorded.
Objective Response Rate as defined by RECIST v1.1. | 60 months
  Objective Response (OR) is defined as achieving a best overall response of complete response (CR) or partial response (PR), as defined using RECIST v1.1. Complete Response (CR): Disappearance of all target lesions. Any pathological lymph nodes (whether target or non-target) must have reduction in short axis to <10 mm. Partial Response (PR): At least a 30% decrease in the sum of diameters of target lesions, taking as reference the baseline sum diameters.
Duration of Disease Control | 60 months
  The Duration of Disease Control is defined as the time from randomization to the date of the first documented disease progression (taking as reference for progressive disease the smallest measurements recorded on study) or death, whichever occurs first.
Adverse events | 60 months
  Adverse events and concomitant medications will be collected throughout the study up to 28 days after the last dose of study treatment. Medical history will be assessed, mutation status will be collected, if available, and an electrocardiogram will be performed at screening. Physical examination, vital signs, and laboratory evaluations will be conducted at screening and throughout the study.
Duration of Objective Response | 60 months
  The evaluation of overall response at each assessment is a composite of target lesion response, non-target lesion response, presence of new lesions.
Disease Control Rate | 60 months
  The disease control rate will be calculated as the total number of patients in each group with best overall response of CR, PR or Stable Disease (SD) divided by the total number of randomized patients in the group and will be compared similarly as Objective Response Rate (ORR.)

CONTACTS AND LOCATIONS:
Locations (82):
- United States (10):
  - Florida Hospital, Orlando, Florida
  - University Cancer Institute, Soynton Beach, Florida
  - Joliet Oncology-Hematology Associates Ltd., Joliet, Illinois
  - Kentucky Cancer Clinic, Hazard, Kentucky
  - Missouri Baptist Cancer Center, St Louis, Missouri
  - Novant Health, Winston-Salem, North Carolina
  - MetroHealth Medical Center, Cleveland, Ohio
  - Center for Biomedical Research LLC, Knoxville, Tennessee
  - Blood and Cancer Center of East Texas, Tyler, Texas
  - Virginia Cancer Specialists PC, Fairfax, Virginia
- Australia (8):
  - Flinders Medical Centre, Bedford Park
  - Austin Health, Heidelberg
  - Royal Hobart Hospital, Hobart
  - St George Hospital, Kogarah
  - Cabrini Hospital Malvern, Malvern
  - Port Macquarie Base Hospital, Port Macquarie
  - Border Medical Oncology, Wodonga
  - The Queen Elizabeth Hospital, Woodville
- Germany (4):
  - Kliniken der Stadt Koln gGmbH, Cologne
  - Asklepios Fachkliniken GmbH, Gauting
  - Martha-Maria Krankenhaus Halle-Dolau gGmbH, Halle
  - Klinikum Kassel, Kassel
- Hungary (4):
  - Orszagos Koranyi TBC es Pulmonologiai Intezet, Budapest
  - Országos Korányi TBC és Pulmonológiai Intézet, Budapest
  - Uzsoki Utcai Korhaz, Budapest
  - Jasz-Nagykun-Szolnok Megyei Hetenyi Geza Korhaz-Rendelointezet, Szolnok
- Israel (2):
  - Meir Medical Center, Kfar Saba
  - Tel Aviv Sourasky Medical Center, Tel Aviv
- Italy (9):
  - Az. Osp. Univ. Ospedali Riuniti Umberto I G.M. Lancisi G.Salesi, Ancona
  - Azienda Ospedaliera Papa Giovanni XXIII, Bergamo
  - Azienda Ospedaliera Istituti Ospitalieri, Cremona
  - Istituto Nazionale per la Ricerca sul Cancro, Genova
  - Ospedale Livorno, Livorno
  - Azienda Ospedaliera - Ospedale San Carlo Borromeo, Milan
  - Azienda Ospedaliera Niguarda Ca Granda, Milan
  - Azienda Ospedaliero Universitaria di Parma, Parma
  - IRCCS Policlinico San Matteo, Pavia
- New Zealand (2):
  - Christchurch Hospital, Christchurch
  - Palmerston North Hospital, Palmerston North
- Poland (4):
  - Samodzielny Publiczny Zespol Gruzlicy i Chorob Pluc w Olsztynie, Olsztyn
  - Med-Polonia Sp. z o.o., Poznan
  - Szpital Kliniczny Przemienienia Panskiego Uniwersytetu Medycznego im. K. Marcinkowskiego w Poznaniu, Poznan
  - Specjalistyczny Szpital im. Alfreda Sokolowskiego, Szczecin
- Russia (5):
  - Arkhangelsk Regional Clinical Oncology Dispensary, Arkhangelsk
  - Federal State Institution Medical Radiology Research Center, Obninsk
  - Consorcio Hospitalario Provincial de Castellon, Saint Petersburg
  - Leningrad Regional Clinical Hospital, Saint Petersburg
  - Oncology Centre Number 2, Sochi
- SOC Clinic @ Farrer Park, Singapore, Singapore
- South Korea (7):
  - Kosin University Gospel Hospital, Busan
  - Keimyung University Dongsan Medical Center, Daegu
  - Gachon University Gil Hospital, Incheon
  - Chonnam National University Hwasun Hospital, Jeonnam
  - Seoul National University Bundang Hospital, Seongnam
  - Korea University Anam Hospital, Seoul
  - Samsung Medical Center, Seoul
- Spain (8):
  - Fundacion Hospital de Alcorcon, Alcorcón
  - Hospital del Mar, Barcelona
  - Consorcio Hospitalario Provincial de Castellon, Castellon
  - Hospital Universitario Insular Materno-Infantil de Las Palmas, Las Palmas de Gran Canaria
  - Hospital Universitario La Paz, Madrid
  - Hospital Universitario Puerta de Hierro, Majadahonda-Madrid
  - Corporacio Sanitaria Parc Tauli, Sabadell
  - Hospital Universitario Doctor Peset, Valencia
- Taiwan (5):
  - Changhua Christian Hospital, Changhua
  - China Medical University Hospital, Taichung
  - Taichung Veterans General Hospital, Taichung
  - National Cheng Kung University Hosptial, Tainan
  - Tri-Service General Hospital, Taipei
- Thailand (6):
  - Saraburi Regional Hospital, Changwat Sara Buri
  - Prapokklao Hospital, Chanthaburi
  - Songklanagarind Hospital Prince of Songkla University, Hat Yai, Songkhla
  - Maharat Nakhonratchasima Hospital, Nakhon Ratchasima
  - National Cancer Institute, Phayathai, Bangkok
  - Buddhachinnaraj Hospital, Phisanulok
- Ukraine (7):
  - Municipal Institution Clinical Oncology Dispensary of Dnipropetrovsk Regional Council, Dnipropetrovsk
  - Municipal institution Multifield City Clinical Hospital Numero 4 of Dnipropetrovsk Regional Council, Dnipropetrovsk
  - MIHC Kharkiv Regional Clinical Oncology Center, Kharkiv
  - Ukrainian Medical Stomatological Academy, Poltava
  - Regional Municipal Institution Sumy Regional Clinical Oncology Dispensary, Sumy
  - Uzhgorod Central City Clinical Hospital, Uzhhorod
  - Vinnytsya Regional Clinical Oncology Dispensary, Vinnytsia